CLINICAL TRIAL: NCT04985812
Title: A Multicenter, Double-blind, Placebo-controlled, Randomized, Multiple Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of JNJ-67484703 in Participants With Active Rheumatoid Arthritis
Brief Title: A Study of JNJ-67484703 in Participants With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR109021; 2021-000195-10 (EudraCT Number); 67484703ARA1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-07-06; First posted 2021-08-02 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- JNJ-67484703 (Experimental): Participants will receive multiple doses of JNJ-67484703.
  Interventions: Drug: JNJ-67484703
- Placebo (Placebo Comparator): Participants will receive multiple doses of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-67484703 — Participants will receive JNJ-67484703.
  Arms: JNJ-67484703
Drug: Placebo — Participants will receive placebo to JNJ-67484703.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate safety and tolerability of JNJ-67484703 administrations in participants with active rheumatoid arthritis (RA).

DETAILED DESCRIPTION:
JNJ-67484703 is a humanized immunoglobulin G1 kappa (huIgG1κ) antibody that is being developed as a treatment for systemic autoimmune disorders. The primary hypothesis of this study is that treatment with JNJ-67484703 as compared to placebo will result in a similar tolerability and safety profile, as a measure of participants with abnormalities in vital signs, physical examinations, and laboratory safety tests. This study will be conducted in 3 phases: screening phase (up to 6 weeks), treatment phase (up to 10 weeks), and follow-up phase (up to 14 weeks). The duration of study participation will be approximately 30 weeks. Safety assessment like electrocardiogram (ECG), adverse events will be performed during the study. Efficacy assessment like joint assessments, pain assessments, RA joint pain severity assessment, patient's and physician's global assessment of disease activity, health assessment questionnaires, duration of morning stiffness, functional assessment of chronic illness therapy-fatigue will be performed during the study.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrated an inadequate response to, or loss of response or intolerance to: at least 1 conventional synthetic disease-modifying antirheumatic drug (csDMARD) and/or up to 2 biologic DMARD (bDMARD)/targeted synthetic DMARD (tsDMARD)
* Have C-reactive protein (CRP) greater than or equal to (>=) 0.3 milligrams per deciliter (mg/dL) at screening
* Medically stable on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening
* Have a diagnosis of rheumatoid arthritis (RA) (American College of Rheumatology [ACR]/ European League Against Rheumatism [EULAR] criteria 2010)
* Body weight within the range of 50.0 kilograms (kg) to 120.0 kg, inclusive, and have a body mass index (BMI) of 19.0 kilograms per meter square (kg/m^2) to 32.0 kg/m^2, inclusive
* All women must have a negative highly sensitive serum (beta-human chorionic gonadotropin [beta-hCG]) at screening

Exclusion Criteria:

* Known allergies, hypersensitivity, or intolerance to any biologic medication or excipients of JNJ-67484703
* Has a diagnosed or reported history or current signs or symptoms indicating severe, progressive, or uncontrolled hepatic, renal, cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances
* Have other known inflammatory diseases that might confound the evaluations of benefit from JNJ-67484703 therapy
* Have a history of any clinically significant adverse reaction to murine or chimeric proteins, including, but not limited to, allergic reactions
* Have a history of or currently have felty's syndrome

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-05-18 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Treatment-emergent Adverse Events (TEAEs) | Up to 24 weeks
  An adverse event (AEs) is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. TEAEs are AEs with onset during the treatment phase or that are a consequence of a pre-existing condition that has worsened since baseline.
Percentage of Participants with Treatment-emergent Serious Adverse Events (SAEs) | Up to 24 weeks
  A serious adverse event based on International Council for Harmonization (ICH) and European Union (EU) guidelines on pharmacovigilance for medicinal products for human use is any untoward medical occurrence that at any dose: a) results in death; b) is life-threatening (the participant was at risk of death at the time of the event. It does not refer to an event that hypothetically might have caused death if it were more severe.); c) requires inpatient hospitalization or prolongation of existing hospitalization; d) results in persistent or significant disability/incapacity; e) Is a congenital anomaly/birth defect; f) is a suspected transmission of any infectious agent via a medicinal product.
Percentage of Participants with TEAEs by System Organ Class (SOC) with a Frequency Threshold of 5 Percent (%) or More | Up to 24 weeks
  Percentage of participants with TEAEs by SOC with a frequency threshold of 5% or more by study intervention will be reported. TEAEs are AEs with onset during the treatment phase or that are a consequence of a pre-existing condition that has worsened since baseline.
Percentage of Participants with Abnormalities in Vital Signs | Up to 24 weeks
  Percentage of participants with abnormalities in vital signs (temperature [oral or tympanic], pulse/heart rate, respiratory rate and blood pressure [systolic and diastolic]) will be reported.
Percentage of Participants with Abnormalities in Physical Examination | Up to 24 weeks
  Percentage of participants with abnormalities in physical examination will be reported.
Percentage of Participants with Abnormalities in Laboratory Parameters | Up to 24 weeks
  Percentage of participants with abnormalities in laboratory parameters (hematology, serum chemistry, and urinalysis) will be reported.

SECONDARY OUTCOMES:
Serum Concentration of JNJ-67484703 Over Time | Up to 24 weeks
  Serum concentration of JNJ-67484703 over time will be reported using a validated, specific, and sensitive method.
Percentage of Participants with Antibodies to JNJ-67484703 in Participants Receiving Active Study Intervention | Up to 24 weeks
  Percentage of participants with antibodies to JNJ-67484703 in participants receiving active study intervention will be reported.
Change from Baseline in Disease Activity Index Score 28 using C-reactive Protein (DAS28-CRP) at Week 12 | Baseline, Week 12
  DAS28-CRP is a derived score combining tender joints (28 joints), swollen joints (28 joints), CRP, and patient's global assessment of disease activity (GH). The set of 28 joint count is based on evaluation of the shoulder, elbow, wrist, metacarpophalangeal (MCP)1, MCP2, MCP3, MCP4, MCP5, proximal interphalangeal (PIP)1, PIP2, PIP3, PIP4, PIP5 joints of both the upper right extremity and the upper left extremity as well as the knee joints of lower right and lower left extremities. Scores below 3.2 indicate best disease control and scores above 5.1 indicate worse disease control.
Percentage of Participants Achieving American College of Rheumatology (ACR)20, ACR50, and ACR70 Response | Up to 24 weeks
  ACR responses are presented as numerical measurement of improvement in multiple disease assessment criteria. For example, ACR20 response is defined as percent improvement of 20 or higher from baseline in both swollen joint count (66 joints) and tender joint count (68 joints), combined with a percent improvement of 20 or higher from baseline in 3 of the following 5 assessments: patient's assessment of pain by visual analog scale (VAS), patient's global assessment of disease activity by VAS, physician's global assessment of disease activity by VAS, patient's assessment of physical function measured by health assessment questionnaire-disability index (HAQ-DI, a 20-question instrument assessing 8 functional areas), and CRP. ACR50 and ACR70 are similarly defined except percent improvement threshold from baseline is 50 and 70, respectively.
Percentage of Participants Achieving DAS28-CRP Remission (less than [<] 2.6) at Week 12 | Week 12
  Percentage of participants achieving DAS28-CRP remission < 2.6 at Week 12 will be reported.
Percentage of Participants Achieving DAS28-CRP Low Disease Activity (<=3.2) at Week 12 | Week 12
  Percentage of participants achieving DAS28-CRP low disease activity (defined as DAS28-CRP less than or equal to [<=] 3.2) at week 12 will be reported.
Change in Number of T-lymphocyte Populations in Blood | Up to 24 weeks
  Change in number of T-lymphocytes in blood will be reported. T-lymphocyte populations in blood will be assessed by flow cytometry.
Change in Magnitude and Duration of Cell Surface Expression Level of Receptors | Up to 24 weeks
  Change in magnitude and duration of cell surface expression level of receptors will be assessed by flow cytometry will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (11):
- United States (2):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - GCSP/CIS Orland Park, Orland Park, Illinois
- Arensia Exploratory Medicine, Tbilisi, Georgia
- Hungary (3):
  - Budai Irgalmasrendi Korhaz, Budapest
  - Clinexpert Kft, Gyöngyös
  - CRU Hungary Kft., Kistarcsa
- Arensia Exploratory Medicine, Chisinau, Moldova
- Spain (3):
  - Hosp Univ A Coruna, A Coruña
  - Hosp. Clinico San Carlos, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
- ARENSIA Exploratory Medicine Unit, Kiev, Ukraine

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Ling ITC, Marciniak SJ, Clarke SH, Lakshminarayanan V, Loza MJ, Liva SG, Wang T, Orillion A, Tikhonov I, Noss EH. Safety, tolerability, and efficacy of the PD-1 agonist antibody JNJ-67484703 in adults with active rheumatoid arthritis: results of a multicenter, double-blind, placebo-controlled, randomized, multiple-dose phase Ib study. Ther Adv Musculoskelet Dis. 2025 Oct 21;17:1759720X251385857. doi: 10.1177/1759720X251385857. eCollection 2025. PMID 41146691